CLINICAL TRIAL: NCT02867072
Title: Laparoscopic Versus Open Appendectomy: A Retrospective Cohort Study Assessing Outcomes and Cost-effectiveness
Brief Title: Laparoscopic Versus Open Appendectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Marco Vacante, MD, PhD, University of Catania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01/2004
Record Dates: First submitted 2016-08-08; First posted 2016-08-15 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis

ARMS (2):
- Open appendectomy (Active Comparator): Subjects that underwent open surgery for appendicitis
  Interventions: Procedure: Open appendectomy
- Laparoscopic appendectomy (Active Comparator): Subjects that underwent laparoscopic surgery for appendicitis
  Interventions: Procedure: Laparoscopic appendectomy

INTERVENTIONS:
Procedure: Open appendectomy
  Arms: Open appendectomy
Procedure: Laparoscopic appendectomy
  Arms: Laparoscopic appendectomy

SUMMARY:
Appendectomy is the most common surgical procedure performed in emergency surgery. Because of lack of consensus about the most appropriate technique, appendectomy is still being performed by both open (OA) and laparoscopic (LA) methods. In this retrospective analysis, the investigators aimed to compare the laparoscopic approach and the conventional technique in the treatment of acute appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* acute appendicitis

Exclusion Criteria:

* Pregnant women and patients with severe medical disease (hemodynamic instability, chronic medical or psychiatric illness, cirrhosis, coagulation disorders) requiring intensive care

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 593 (Actual)
Dates: Start 2004-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Hospital cost | 3 days
  Mean hospital cost (in Euro) for patients that underwent appendectomy
Wound infection | 1 week
  Number of patients with wound infection after appendectomy

REFERENCES:
- [Derived] Biondi A, Di Stefano C, Ferrara F, Bellia A, Vacante M, Piazza L. Laparoscopic versus open appendectomy: a retrospective cohort study assessing outcomes and cost-effectiveness. World J Emerg Surg. 2016 Aug 30;11(1):44. doi: 10.1186/s13017-016-0102-5. eCollection 2016. PMID 27582784